CLINICAL TRIAL: NCT04206709
Title: Influence of Single Session of Aerobic Exercise on Acute Pain and Function in Patients After Total Knee Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Haifa (Other)
Collaborators: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2019-07-04; First posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-07

CONDITIONS: Total Knee Replacement
Keywords: exercise induced analgesia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic effort (Experimental): Active upper limbs pedaling
  Interventions: Procedure: aerobic effort
- passive pedaling (Sham Comparator): passive pedaling
  Interventions: Other: passive pedaling

INTERVENTIONS:
Procedure: aerobic effort — Active upper limbs pedaling while maintaining a pulse calculated to be approximately 60% of the predicted maximum heart rate of each patient for 20 minutes.
  Arms: aerobic effort
Other: passive pedaling — 20 minutes passive pedaling by upper limbs.
  Arms: passive pedaling

SUMMARY:
The purpose of this study is to examine the immediate effect of aerobic exercise effort on clinical and experimental pain, knee active range of motion and function in people after total knee replacement.

DETAILED DESCRIPTION:
Total knee replacement is a prevalent orthopedic elective surgery in the Western world. After surgery, especially in the first two weeks, patients suffer from high degrees of pain that may lead to delayed recovery, increased risk to chronic pain and pain comorbidities, and may harm the knee function. In purpose to alleviate the pain, most patients tend to passive coping strategies which include the use of high levels of analgesics, including steroids, which may have accompanying side effects.

Aerobic activity is found to have a beneficial effect on pain threshold and pain tolerance in healthy subjects and in chronic pain syndromes. Researches indicate that single bout of aerobic effort increase pain threshold and pain tolerance and decrease pain severity for 15-30 minutes. Until now, the effect of a one-time aerobic effort has not been tested on subjects suffering from acute pain following surgical intervention.

This trail will examine the immediate effect of single aerobic effort on clinical and experimental pain, active knee range of motion and function among people with acute pain after total knee replacement.

40 subjects undergoing total knee replacement at the medical Center for Galilee as a result of Osteoarthritis in one of they knee, will be recruited to the study. The study will take place during the hospitalization in the 5th and 6th days after surgery. In those 2 days the subjects will participate in two meetings: in one session, the participants will be asked to perform active pedaling for 20 minutes in their upper limbs of a pulse that will be calculated approximately 60% of their maximum predictive pulse. in the second meeting the participants will perform passive training with their upper limbs for the same duration. The order of interventions will be randomly determined. Before and after the intervention, it will be examined by pain measures (pressure pain threshold, spontaneous pain perception and arousal pain by the Visual Analogue Scale (VAS) scale), at rest, in a sitting-standing-sitting transfers, while carrying an equal weight on both feet and while walking. the active range of motion of the operated knee, and functional measures - 10 Meters walk Test and Timed Up and Go test.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for unilateral total knee replacement surgery in the Department of Orthopedics 'A", at f the Galilee Medical Center.
* 18 years and older.
* Diagnosed with osteoarthritis.
* Consent to participate in the trial.
* Understand simple instructions.
* Capable of walking with walking aid independently or supervised.
* Allowed to perform medium-intensity aerobic exercise to-60% of their predicted maximum pulse.

Exclusion Criteria:

* Individuals who have a physical limitation preventing them from performing active pedaling in upper limbs for 20 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Pressure Pain Threshold (PPT) | Change from Baseline PPT will be assessed right after the intervention
  PPT examination by designated device
Visual Analogue Scale (VAS) | Change from Baseline VAS will be assessed right after the intervention
  100mm VAS -A vertical VAS ruler with a slider indicator and a scale of 0-100 mm on the ruler's front side was used. the lower edge marked "0" and the upper edge marked "100". The back side of the ruler included a "happy" face figure at the lower edge representing "no pain" and a "sad" face at the upper edge representing "severe pain". Higher VAS scores equal more pain.
10 Meter Walk Test | Change from 10 meter walk test baseline outcome will be assessed right after the intervention
  timed 10 meter walk test

SECONDARY OUTCOMES:
Knee Active Range of Motion (aROM) | Change in aROM baseline will be assessed right after the intervention
  Goniometer measure
Timed Up and Go (TUG) | Change from TUG test outcome will be assessed right after the intervention
  Timed Up and Go test

CONTACTS AND LOCATIONS:
Overall Officials: Einat Kodesh, PhD, Principal Investigator — University of Haifa; Noa Katz-Betzalel, Study Director — Galilee Medical Center
Locations (1):
- Galilee Medical Center, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: No